CLINICAL TRIAL: NCT06739369
Title: Investigation of the Relationship Between Arterial Stiffness and Pulmonary and Extrapulmonary Features in Patients With Ankylosing Spondylitis
Brief Title: The Relationship Between Arterial Stiffness and Pulmonary and Extrapulmonary Features in Ankylosing Spondylitis
Status: Recruiting | Type: Observational
Sponsor: Kirsehir Ahi Evran Universitesi (Other)
Responsible Party: Principal Investigator, Merve Firat, Assistant Professor, Kirsehir Ahi Evran Universitesi
Other Study IDs: 2024-14/120
Record Dates: First submitted 2024-11-27; First posted 2024-12-18 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2024-11

CONDITIONS: Ankylosing Spondylitis (AS)
MeSH Terms: conditions — Spondylitis, Ankylosing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Ankylosing spondylitis

SUMMARY:
The aim of this study was to investigate the relationship between arterial stiffness and pulmonary and extrapulmonary features in patients with ankylosing spondylitis.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ankylosing spondylitis according to ASAS diagnostic criteria
* Being aged 18-65
* Stable medication use for at least 3 months
* Voluntary participation in the study

Exclusion Criteria:

* Having uncontrolled cardiopulmonary disease
* Being pregnant
* Having undergone recent surgery
* Presence of malignancy
* Failure to perform to assessments

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients followed up with a diagnosis of ankylosing spondylitis will be included.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-08-06 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Arterial stiffness | 1st day
  It will be evaluated with brachial pulse waves.
Respiratory muscle strength | 1st day
  Maximal inspiratory pressure (MIP) and maximal expiratory pressure (MEP) will be measured using a portable mouth pressure device.
Respiratory muscle endurance | 1st day
  This will be evaluated with increased workload testing.
Exercise capacity | 1st day
  Exercise capacity will be assessed with 6 minute walk test.
Peripheral muscle strength | 1st day
  Hand grip strength will be assessed with a grip dynamometer.
Muscle function | 1st day
  It will be evaluated with one-minute sit to stand test

SECONDARY OUTCOMES:
Physical activity | 1st day
  Physical activity level will be evaluated using International Physical Activity Questionnaire-Short form
Forced vital capacity | 1st day
  Forced vital capacity (FVC) will be assessed using spirometry.
Forced expiratory volume in one second | 1st day
  Forced expiratory volume in one second (FEV1) will be assessed using spirometry.
Forced expiratory volume in one second/forced vital capacity ratio | 1st day
  Forced expiratory volume in one second/forced vital capacity ratio will be assessed using spirometry.
Peak expiratory flow | 1st day
  Peak expiratory flow (PEF) will be assessed using spirometry.
Forced mid-expiratory flow | 1st day
  Forced mid-expiratory flow (FEF25-75) will be assessed using spirometry.

CONTACTS AND LOCATIONS:
Locations (1):
- Kirsehir Ahi Evran University, Kırşehir, Turkey (Türkiye)